CLINICAL TRIAL: NCT05588180
Title: Comparing The Ratio Of Femoral Vein Diameter To Femoral Artery Diameter With Pulse Pressure Variation As A Diagnostic Tool For Fluid Responsiveness In Mechanically Ventilated Patients; A Prospective Observational Study
Brief Title: The Ratio Of Femoral Vein Diameter To Femoral Artery Diameter With Pulse Pressure Variation As A Diagnostic Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, ASSOCIATE PROFESSOR OF ANESTHESIA, Fayoum University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: M 600
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Mechanically Ventilated Patients
Keywords: mechanically ventilated patients; FVD / FAD

STUDY DESIGN:
Intervention Model Description: group (F) FVD/FAD ratio guided
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (P) (Active Comparator): Group (P) PPV guided group
  Interventions: Procedure: PPV
- Group (F) (Active Comparator): Group (F) FVD/FAD ratio guided
  Interventions: Procedure: FVD/FAD ratio guided

INTERVENTIONS:
Procedure: FVD/FAD ratio guided — Ultrasound-guided ratio
  Arms: Group (F)
Procedure: PPV — PPV
  Arms: Group (P)

SUMMARY:
In assessing critically ill patients, an accurate assessment of a patient's volume status and whether they will respond to a fluid challenge with an increase in cardiac output is vital. 1 When hypovolemia is detected, volume expansion is utilized to enhance hemodynamics and restore normal blood pressure. 2 Hemodynamic tests (right atrial pressure, pulmonary artery occlusion pressure, and cardiac output ) are used to assess preload in critically ill patients, although these indexes are not necessarily reliable predictors of fluid status. According to the Starling law, fluid administration is hypothesized to boost cardiac output by raising preload, which describes a positive relationship between cardiac muscle fiber length and contractility. However, the Starling curve hits a plateau beyond its ascending leg, and additional fluid administration can be hazardous, leading to right ventricular overload and pulmonary edema Invasive or noninvasive techniques can be used to determine blood volume status. Assessments such as central venous pressure (CVP) and mean pulmonary artery pressure (mPAP) are both invasive procedures. Various factors influence CVP (including thoracic, pericardial, abdominal pressures, etc.). CVP can be used as a fluid management indication, although It can be misused to estimate blood volume or mislead methods for treatment. Dynamic indices such as stroke volume variation (SVV) and pulse pressure variation (PPV) are superior to static indices for assessing volume status. However, these dynamic indices are unreliable when a patient is ventilated with low tidal volume, such as acute respiratory distress syndrome (ARDS); the tidal volume is insufficient to change intrathoracic pressure significantly. Ultrasound (US) evaluation of the inferior vena cava (IVC) may help determine fluid status.

DETAILED DESCRIPTION:
The study will be conducted in intensive care units of Fayoum University Hospitals after approval of the local institutional ethics committee, and the local institutional review board will approve the study. The inclusion criteria will be as follows: patients on mechanical ventilation(MV), aged between 18 and 60 years with circulatory failure defined as mean arterial pressure (MAP) less than 65 mmHg or systolic arterial pressure less than 90mm Hg with signs of hypoperfusion (urinary flow < 0.5mL/kg/ min for > 2hr, tachycardia > 100 beats/min, or presence of skin mottling, and serum lactate more than 2 mmol/L) 17 and showing positive PLRT. The exclusion criteria: cardiac arrhythmias, previously known significant valvular disease or intracardiac shunt, air leakage through chest drains, increasing intraabdominal pressure, norepinephrine infusion as it decreases PPV and SVV, masking their ability for the detection of FR15

, peripheral vascular diseases, ARDS patients due to low tidal volume a, Contraindication for fluid administration as cardiogenic shock, acute pulmonary edema or LVEF% less than 50%. , renal patients with oliguria and volume overload including patients on hemodialysis or patients with acute anuric renal failure., patients with lower extremity artery/vein thrombosis, significant lower extremity artery plaque, lower extremity artery occlusion, inferior vena cava filter implantation, lower extremity varicose veins,

All patients fulfilling criteria will be monitored by (1) 6 leads ECG, (2) noninvasive BP, (3)urinary catheter for UOP, (4) pulse oximeter then divided into 2 groups, group (P) PPV guided group and group (F) FVD/FAD ratio guided

Randomization of patients to each of the treatment groups will be done by a statistician not involved in the study, using the website randomization.com. The allocation concealment will be done by contacting the statistician giving him the patient number, age, and sex to receive the patient allocation in a sealed envelop.

The envelope is to be received and opened after the informed consent is obtained Neither the participants, the study investigator, the attending clinicians, nor the data collector will be aware of groups allocation till the study end. The Consolidated Standards of Reporting Trials (CONSORT)recommendation will be followed. Group (P):(n=30), patients will be temporarily sedated and paralyzed and on fully controlled mechanical ventilation. No spontaneous breathing effort will be detected on the mechanical ventilator waveform monitor, ensuring that the respiratory changes in arterial pressure reflect only the effects of positive pressure ventilation. Modes of ventilation are selected to volume or pressure-controlled ventilation, depending on the decision of the primary physicians. A tidal volume will be set to not less than 8 ml/ kg (predicted body weight). The preset respiratory rate will be set at 14 breaths/min. Positive end-expiratory pressure (PEEP) will be between 8 and 10 cmH2O. The plateau pressure was kept at below 30 cmH2O. In all patients, radial artery cannulation will be done for invasive blood pressure monitoring (using a 20 G cannula), PPV is calculated directly on Nihon Kohden monitors at the base line then infusion of 4ml/kg /h of crystalloids will be infused till PPV will be less than 13%. 15

Group(F) : (n=30), FVD/FAD ratio guided; US probe will be used first to find the bifurcation position of the femoral artery, and then the probe will be retracted proximally. The visual field of the bifurcation will disappear until the probe enters the main branch of the femoral artery, and the femoral artery and vein could be observed simultaneously. Under normal conditions, pulsation indicates the femoral artery, and its companion is the femoral vein. The mean FVD and FAD will be measured then the FVD / FAD ratio will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* patients on mechanical ventilation

Exclusion Criteria:

* cardiac arrhythmias
* previously known significant valvular disease or intracardiac shunt
* air leakage through chest drains
* increasing intraabdominal pressure
* norepinephrine infusion as it decreases PPV and SVV
* peripheral vascular diseases
* ARDS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
MAP | the first 48 hours postoperative
  mean arterial blood pressure

SECONDARY OUTCOMES:
the cutoff value of FVD/FAD reflecting FR | the first 48 hours postoperative
  the cutoff value of FVD/FAD reflecting FR
PPV | the first 48 hours postoperative
  pulse variation index

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamed, M D, Principal Investigator — Fayoum University Hospital
Locations (1):
- Fayoum University hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Result] Kalantari K, Chang JN, Ronco C, Rosner MH. Assessment of intravascular volume status and volume responsiveness in critically ill patients. Kidney Int. 2013 Jun;83(6):1017-28. doi: 10.1038/ki.2012.424. Epub 2013 Jan 9. PMID 23302716
- [Result] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374